CLINICAL TRIAL: NCT06374186
Title: COntinuous Glucose Monitoring, Contingency Management, and Motivational InTerviewing for Patients With TypE 2 Diabetes in Kansas City
Acronym: COMMITTED2-KC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri, Kansas City (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2095072; 2095072 (Other: UMKC IRB)
Record Dates: First submitted 2024-04-15; First posted 2024-04-18 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 Diabetes; Glucose; contingency management; motivational interviewing
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Behavior Therapy; Motivational Interviewing

STUDY DESIGN:
Intervention Model Description: A randomized parallel-group pilot study of a combination intervention using Motivational Interviewing (MI) and Contingency Management (CM) for patients with T2DM.
Who Masked: Care Provider
Masking Description: Because this is a behavioral intervention, participant blinding is not possible. Randomization will occur after baseline assessment and participants will be instructed to not tell their provider their assigned condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behavioral Intervention with financial rewards and coaching (Experimental): Individuals in the treatment group will receive financial rewards (contingency management) and diabetes coaching (motivational interviewing) in addition to wearing a continuous glucose monitor while receiving their usual diabetes treatment.
  Interventions: Behavioral: Behavioral Intervention with financial rewards and coaching
- Control (Active Comparator): Individuals in the control group will not receive any interventions and will only wear a continuous glucose monitor while receiving their usual diabetes treatment.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Behavioral Intervention with financial rewards and coaching — Participants will receive variable financial incentives based on their engagement with the continuous glucose monitor and meeting diabetes treatment goals. In addition, they will participate in three motivational interviewing sessions focused on their diabetes management. Participants will continue to receive their diabetes treatment as usual.
  Other Names: Contingency management and motivational interviewing
  Arms: Behavioral Intervention with financial rewards and coaching
Behavioral: Control — Participants will only receive a continuous glucose monitor, which they may engage with as desired and no further intervention. Participants in the control group will continue to receive their diabetes treatment as usual.
  Arms: Control

SUMMARY:
This study is evaluating a behavioral treatment program that uses diabetes coaching and financial rewards in addition to continuous glucose monitoring to improve diabetes management in adult patients with type 2 diabetes. This study will evaluate if this behavioral treatment program increases individual adherence to a diabetes treatment plan and improves blood sugar management.

DETAILED DESCRIPTION:
A randomized parallel-group pilot study of a combination intervention using Motivational Interviewing (MI) and Contingency Management (CM) for patients with T2DM. Individuals will be randomized in a 1:1 ratio to the intervention group or the control group. Randomization will be blocked and stratified by long-acting insulin and GLP1 medication use. All participants will be given a Continuous Glucose Monitor (CGM) to assess real-time blood sugar levels and establish CM rewards for those assigned to the treatment group.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with type 2 diabetes
2. Age 18 to 65
3. Hemoglobin A1c (blood draw or point-of-care) test available within the last 3 months
4. Most recent hemoglobin A1c result between 8.0 and 11.0
5. Currently receiving treatment for diabetes by a licensed healthcare provider.
6. Reliable access to a personal smart phone that is compatible with CGM
7. English speaking

Exclusion Criteria:

1. Type 1 diabetes
2. Secondary type 2 diabetes (diagnosis secondary to other medical conditions such as pancreatitis, Cystic Fibrosis, or Cushing disease)
3. Prescribed short-acting (mealtime) insulin as part of diabetes treatment plan
4. Known or acknowledged active substance use disorder or that would interfere or negatively impact participation in the study
5. Diagnosis of a medical/psychiatric condition that would prevent participation in the study (e.g., Intellectual Disability, Alzheimer's disease, Traumatic Brain Injury, Schizophrenia)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-07-29 (Actual); Study Completion 2025-08-12 (Actual)

PRIMARY OUTCOMES:
Time in target blood glucose range per CGM | baseline to 14 weeks
  Percent time with blood glucose between 70 to 180 mg/dL
Hemoglobin A1C | baseline to 12 weeks
  laboratory value

SECONDARY OUTCOMES:
Diabetes Quality of Life Brief Inventory | baseline to 12 weeks
  self-report questionnaire
Diabetes Distress Scale | Baseline to 12 weeks
  self-report questionnaire
PROMIS Medication Adherence Scale | Baseline to 12 weeks
  self-report questionnaire
Perceived Dietary Adherence Questionnaire | Baseline to 12 weeks
  self-report questionnaire
Motivation and Confidence Ruler | Baseline to 12 weeks
  self-report questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Jared Bruce, PhD, Principal Investigator — University of Missouri, Kansas City
Locations (1):
- University of Missouri - Kansas City School of Medicine, Kansas City, Missouri, United States